CLINICAL TRIAL: NCT03789084
Title: A Hybrid Type 1 Trial Evaluating the Feasibility, Acceptability, Preliminary Effectiveness of Brief Cognitive-behavioral Therapy for Health Anxiety Delivered by Medical Assistants in Primary Care
Brief Title: Hybrid Trial of Brief Cognitive-Behavioral Therapy for Health Anxiety in Primary Care
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dartmouth-Hitchcock Medical Center (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Robert E. Brady, Assistant Professor, Dartmouth-Hitchcock Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: D19044; 6K23MH116367-02 (NIH)
Record Dates: First submitted 2018-12-26; First posted 2018-12-28 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2026-01

CONDITIONS: Illness Anxiety Disorder; Somatic Symptom Disorder; Health Anxiety

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cognitive-Behavioral Therapy (Experimental): Brief Cognitive-Behavioral Therapy for Health Anxiety
  Interventions: Behavioral: Brief Cognitive-Behavioral Therapy for Health Anxiety
- Referral to mental health provider (Other): Provider makes referral to a mental health provider
  Interventions: Behavioral: Referral to mental health provider

INTERVENTIONS:
Behavioral: Brief Cognitive-Behavioral Therapy for Health Anxiety — 4-session in-person 45-minute psychotherapy sessions focused on building motivation for change, psychoeducation, cognitive restructuring, and situational and interoceptive exposure to health-related fear stimuli.
  Arms: Cognitive-Behavioral Therapy
Behavioral: Referral to mental health provider — Provider makes a referral to a mental health provider in the outpatient psychiatry clinic or a community provider of the participant's choice.
  Arms: Referral to mental health provider

SUMMARY:
This study is a randomized controlled pilot trial using a hybrid type 1 effectiveness-implementation design to evaluate the feasibility, acceptability, and preliminary effectiveness of a brief cognitive-behavioral intervention delivered by medical assistants in a primary care setting. The trial compares clinical outcomes of participants assigned to the intervention condition to those of participants assigned to a usual care condition. The clinical outcome is change on a self-report measure of health anxiety. Assessments occur at baseline, four weeks, and 12 weeks post-treatment. The study will also measure engagement with the intervention and assess feasibility and acceptability of the intervention in terms of fidelity of trained study therapists and ratings of the intervention by participants. The usual care condition consists of a referral to a mental health provider. The intervention is comprised of four sessions of individually administered cognitive-behavioral therapy addressing health anxiety. Treatment focuses on building motivation for change, psychoeducation about health anxiety, cognitive restructuring, and situational and interoceptive exposure. The study will recruit from three primary care clinics within the Dartmouth-Hitchcock Health system. The study will also assess facilitators and barriers to implementation using qualitative analyses of interview responses provided by the medical assistants delivering the intervention, primary care providers, and clinic administrators at the study sites.

DETAILED DESCRIPTION:
Seventy-two health anxious patients with a diagnosis of Illness Anxiety Disorder or Somatic Symptom Disorder will be randomly assigned to either receive brief cognitive-behavioral therapy (CBT) administered by a medical assistant in the primary care practice where the patient receives their primary care services (intervention condition) or receive a referral to a mental health provider within the outpatient psychiatry clinic or another community provider of their choice (usual care condition). Randomization will be determined by a random number generation program at the point of enrollment. The randomization scheme will be stratified by primary care site to reduce site effects. The primary care sites from which patients will be recruited include the General Internal Medicine clinic at Dartmouth-Hitchcock Medical Center, Dartmouth-Hitchcock Heater Road clinic, and Dartmouth-Hitchcock Manchester. Recruitment will be evenly distributed across sites. The investigators will over-sample racial and ethnic minority patients at Dartmouth-Hitchcock Manchester due to the higher proportion of minority patients receiving services at that location.

The brief CBT intervention is a 4-session psychotherapy comprised of techniques guided by cognitive-behavioral theory and specifically derived from previously published materials. Each technique has support from prior randomized controlled trials demonstrating their efficacy for reducing symptoms of health anxiety and expert consensus. The techniques employed include motivational interviewing, psychoeducation, cognitive restructuring, and situational and interoceptive exposure. Each session of brief CBT is 45-minutes in duration and is delivered by a medical assistant who is principally located at the patient's primary care practice. All sessions are based on a manual developed by the Principal Investigator that includes essential elements to deliver at each session, scripts to guide delivery of the intervention, and homework assignments for the patient to complete between sessions and after completion of the final session. The Principal Investigator provides clinical supervision of the intervention over the course of the study.

The referral process employed in the usual care condition consists of an electronic referral made by the patient's primary care provider to a mental health provider within the Dartmouth-Hitchcock Health system, or a community provider outside of the system identified by the patient in consultation with the primary care provider. The nature of the intervention provided by the mental health provider is not prescribed or guided by the study protocol.

Examination of distributions of all variables using descriptive analyses will precede inferential statistical analysis. Transformations or recoding will be applied to normalize continuous data when necessary. The success of random assignment will be evaluated by comparing the two study groups on baseline characteristics using chi-square tests for categorical variables and t-tests for continuous covariates. If baseline variables are significantly different between groups and are significantly associated with the outcomes (e.g., medical comorbidity), the investigators will include them as covariates in the analytic models.

The primary outcome of change in health anxiety will be tested using a model that accommodates attrition and is appropriate for correlated data due to clustering (by 3 sites and 6 medical assistants) and repeated measures (baseline, 4 and 12 weeks) on the outcomes. Because there are only three assessment points, time will be treated as discrete and fitted to a covariance pattern model to compare average change between groups over time. Group (CBT vs usual care), time (baseline, 4 and 12 weeks), and the group by time interaction will be specified for the model. The treatment effect of intervention relative to control will be evaluated by testing significance of the group by time interaction term. An unstructured variance-covariance structure will be specified to account for the correlated nature of the data due to repeated measures.

The cluster size at site and provider levels are too small to be treated as random effects; therefore, the analysis will take clustering effects due to site and provider into account using small-sample robust estimate correction options implemented in the Statistical Analysis Software (SAS) generalized linear mixed models procedure (PROC GLIMMIX) procedure. GLIMMIX facilitates conducting mixed-effects and generalized estimating equation (GEE) modeling in the same procedure simultaneously.

The sample size was determined by a combination of recruitment feasibility, study therapist (medical assistant) availability, and power analysis. Given two groups, 3-assessment points, and sample size of 72 (36 per arm) with 15% attrition at 12 months (N = 58), and assuming cross-time correlation of 0.60, alpha of 0.05, and two-tailed tests, the study achieves 80% power to detect a minimum effect size of 0.69, between medium (0.50) and large (0.80) in Cohen's d-metric. If the analysis takes clustering effects due to site and providers into account by adjusting the sample size with an intraclass correlation (ICC) of 0.01, the study achieves 80% power to detect an effect size of 0.72. Statisticians recommend ICC between 0.01 and 0.02 in clinical studies with clustering; the investigators used ICC = 0.01 for this power calculation. A larger sample size is needed to detect effect sizes smaller than 0.69 and 0.72; however, sample size for pilot study should be based on pragmatics of recruitment and the necessities for examining feasibility, and not for purpose of inferential statistical tests.

The investigators will assess acceptability of the intervention and strategy using scores on a self-report measure of treatment acceptability using mean scores above a predetermined cut score denoting moderate acceptability across all participants. The investigators assess study therapist fidelity to the treatment by compiling standardized fidelity ratings for each session, nested within each provider, and converted to a percentage fidelity score.

Finally, the investigators will assess acceptability qualitatively using qualitative interviews with medical assistants, primary care providers, and clinic administrators. Interview data will be transcribed and entered verbatim into a qualitative data management software package for content analysis. Content analysis consists of reviewing the responses of interviewees to identify responses that are coded to correspond to Consolidated Framework for Implementation Research constructs. Coding will be conducted by two independent coders (the Principal Investigator and a research assistant) and overseen by a medical anthropologist.

ELIGIBILITY:
Inclusion Criteria:

* Age of 18 years to 85
* Have a primary care provider at Dartmouth-Hitchcock Medical Center-General Internal Medicine, Dartmouth-Hitchcock Heater Road Clinic, or Dartmouth-Hitchcock Manchester
* Primary care visit frequency of two standard deviations above the mean for patients in the individual's age by gender cohort
* Elevated self-reported health anxiety (≥2 on Whiteley Index-7)
* Diagnosis of illness anxiety disorder or somatic symptom disorder determined by Health Anxiety Interview

Exclusion Criteria:

* Non-English speaking
* Chronic medical illness necessitating an increased visit frequency confirmed through consultation with the patient's primary care provider
* Active suicidal ideation
* Unmanaged psychosis or unmanaged bipolar disorder

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Actual)
Dates: Start 2019-03-26 (Actual); Primary Completion 2025-07-01 (Actual); Study Completion 2025-10-30 (Actual)

PRIMARY OUTCOMES:
Change from baseline in health anxiety, measured by the Short Health Anxiety Inventory | Baseline, Post-treatment (4 weeks followup), 12-weeks Post-Treatment (12 weeks followup)
  The Short Health Anxiety Inventory is an 18-item measure of health anxiety in which respondents identify which statement applies best to them among four choices per item scored from 0 to 3 (e.g., "I do not worry about my health" = 0, "I spend most of my time worrying about my health" = 3). The scale range is 0 to 54. Higher scores correspond to increased health anxiety.

SECONDARY OUTCOMES:
Acceptability of the intervention, measured by the Treatment Evaluation Inventory-Short Form | Post-treatment (4 weeks followup), 12-weeks Post-Treatment (12 weeks followup)
  The Treatment Evaluation Inventory-Short Form is a 9-item measure of treatment acceptability (e.g., "I like the procedures used in this treatment") rated on a five-point Likert scale from "strongly disagree" to "strongly agree" and modified to focus on interventions administered to adults. The scale range is 9 to 45. Higher scores correspond to greater acceptability of the intervention.
Change in readiness for intervention, measured by the University of Rhode Island Change Assessment-Psychotherapy Version | Baseline, Post-treatment (4 weeks followup), 12-weeks Post-Treatment (12 weeks followup)
  The University of Rhode Island Change Assessment-Psychotherapy Version is a 32-item measure of readiness for change. Items are rated on a five-point Likert scale from "strongly disagree" to "strongly agree" for each item (e.g., "I think I might be ready for some self-improvement."). The scale range is 32 to 160. Higher scores correspond to increased readiness for change.

OTHER OUTCOMES:
Fidelity to the intervention following training, measured by the Cognitive Therapy Scale-Revised | 1 to 15 months before Baseline
  The Revised-Cognitive Therapy Scale is a 12-item measure of therapist fidelity to cognitive-behavioral therapy (CBT). Items are rated on a seven-point scale of ability to apply CBT principles (0 = "Incompetent" to 6 = "Expert"), by an evaluator with expertise in CBT. A score of ≥36 is the recommended cut-off for CBT fidelity. The scale range is 0 to 72. Higher scores correspond to greater fidelity to the CBT model.
Psychiatric diagnostic comorbidity, assessed by the Mini-International Neuropsychiatric Interview | Baseline
  The Mini-International Neuropsychiatric Interview (MINI) is a widely used brief structured psychiatric diagnostic interview for 17 International Classification of Diseases-10 psychiatric disorders. Each item from the MINI is answered in a dichotomous, yes/no format with additional prompts used by the assessor to clarify ambiguous responses.
Medical diagnostic comorbidity, assessed by the Charlton Age-Comorbidity Index | Baseline
  The Charlson Age-Comorbidity Index is a combined age and comorbidity index in which each decade of life ≥50 years equals a 1-point increase in comorbidity alongside scores assigned to specific disease states. Scores range from 0 to 39, with comorbidities of greater severity assigned higher scores of 1, 2, 3, or 6. Higher scores are associated with greater likelihood of death from the identified comorbid conditions.
Determination of health anxiety diagnoses, assessed by the Health Anxiety Interview | Baseline
  The Health Anxiety Interview (HAI) is a brief clinician-administered semi-structured interview of health anxiety and related disorders. The HAI can be administered in approximately 30 minutes. Reliability data are not available for the HAI, but it has been used successfully in health anxiety outcome trials research. The HAI will be used to verify the presence of excessive health anxiety identified on the WI-7.
Measurement of health anxiety for screening purposes, assessed by the Whiteley Index-7 | 1 week to 1 month before Baseline
  The Whiteley Index-7 (WI-7) is comprised of seven items assessing health anxiety. Respondents indicate how much an item is representative of them (e.g., "Do you often worry about the possibility that you have a serious illness'') using dichotomous scaling. The WI-7 has good sensitivity and specificity for identification of excessive health anxiety. A score of ≥2 is indicative of excessive health anxiety. The scale range is 0 to 7. Higher scores correspond to greater health anxiety.

CONTACTS AND LOCATIONS:
Overall Officials: Robert E Brady, PhD, Principal Investigator — Dartmouth-Hitchcock Medical Center
Locations (1):
- Dartmouth-Hitchcock Medical Center, Lebanon, New Hampshire, United States

IPD SHARING:
Plan to Share IPD: Yes
Study results will be posted to ClinicalTrials.gov in a timely manner with the goal of posting the results as soon as possible following completion of primary analyses and not more than one year after completion of the final participant's participation in the trial. This corresponds to the third year of the career development award period for the hybrid trial covered in this study record. Deidentified individual participant data (IPD) will be available upon request from researchers with a sound research and analytic plan, including replication or inclusion in meta-analysis. IPD will be available immediately and indefinitely following primary outcome manuscript publication.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: IPD will be available immediately and indefinitely following primary outcome manuscript publication.
Access Criteria: Replication trials, meta-analyses; requests should be made directly to Principal investigator at Robert.E.Brady@hitchcock.org.

REFERENCES:
- [Background] Brady RE, Hegel MT, Curran GM, Asmundson GJG, Xie H, Bruce ML. Evaluation of a brief psychosocial intervention for health anxiety delivered by medical assistants in primary care: Study protocol for a pilot hybrid trial. Contemp Clin Trials. 2021 Dec;111:106574. doi: 10.1016/j.cct.2021.106574. Epub 2021 Oct 7. PMID 34628077
- [Background] Brady RE, Braz AN. Challenging Interactions Between Patients With Severe Health Anxiety and the Healthcare System: A Qualitative Investigation. J Prim Care Community Health. 2023 Jan-Dec;14:21501319231214876. doi: 10.1177/21501319231214876. PMID 38041442